CLINICAL TRIAL: NCT00946218
Title: Diagnosis and Characterization of Dengue Fever in Children
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DENGEN
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Part A: Children with presumptive dengue infection enrolled for empiric cost modeling with retrospective clinical estimation and comparison of test performance to the standard of care.
- Part B: Children with definitive dengue infection enrolled for gene expression analysis.

SUMMARY:
Dengue virus is an arbovirus transmitted by mosquitoes which causes significant morbidity and mortality among children in tropical regions, especially in resource limited countries. The objective of this protocol is to compare the sensitivity and specificity of clinical gestalt and two rapid antigen tests for dengue virus and to compare the gene expression of leukocytes in distinct dengue fever disease phenotypes module-based RNA microarray technology.

DETAILED DESCRIPTION:
This is a biology protocol with no treatment regimen associated. Blood collection will be drawn from subjects in El Salvador to be tested in an effort to improve detection and test sensitivity and specificity of a dengue NS1 Ag ELISA, dengue NS1 Ag STRIP, and clinical suspicion for the detection of dengue virus infection in children in San Salvador, El Salvador compared to the gold standard, PCR. This protocol will also seek to identify and compare gene transcription patterns characteristics of each dengue virus disease phenotype in children.

ELIGIBILITY:
Inclusion Criteria Part A:

* Age: Greater than or equal to 6 months and less than 13 years
* One of the following; History of fever OR a history of spontaneous or provoked bleeding

Inclusion Criteria Part B:

* Gender: Female
* Age: greater than or equal to 36 months
* Tanner stage less than 2
* One of the following criteria: Classical Dengue Fever, Dengue Hemorrhagic Fever or Dengue Shock Syndrome

Exclusion Criteria for both parts:

* Obvious alternative explanation for the actual illness
* Cellulitis/Abscess
* Osteomyelitis
* Varicella
* Urinary Tract Infection
* Known immunocompromising condition

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children subject presenting to Benjamin Bloom Children's Hospital in San Salvador, El Salvador.
Sampling Method: Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To compare the sensitivity of dengue NS1 (influenze protein) Ag Enzyme-linked Immunosorbent Assay and dengue NS1 Ag STRIP and WHO clinical diagnostic criteria when applied to children in El Salvador. | 1 year

SECONDARY OUTCOMES:
To identify differences in host leukocyte gene expression in children with DF, DHF, and DSS using high throughput gene expression arrays. | 1 Year
To develop a clinical risk algorithm for predicting severe dengue using NS1 Ag testing techniques and clinical data. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Adderson, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States
- Hospital Nacional de Ninos Benjamin Bloom, San Salvador, El Salvador, El Salvador

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org